CLINICAL TRIAL: NCT03905616
Title: Hierarchical Processing of Visual Movement
Brief Title: HIERARCHY OF VISION
Acronym: HIERARCHY
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: abandonment
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL18_0933; 2019-A00465-52 (Other: ID-RCB)
Record Dates: First submitted 2019-04-04; First posted 2019-04-05 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Neurologic Signs
Keywords: Vision; perception; BOLD activity
MeSH Terms: conditions — Neurologic Manifestations | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- healthy subjects (Experimental): 25 healthy subjects with a normal/corrected vision fitting to all of the inclusion/exclusion criteria. All the subjects will be tested on the same visual stimuli, leading to intrasubject comparison analyses of functional magnetic resonance imaging (fMRI) activity between conditions.
  Interventions: Device: functional Magnetic Resonance Imaging

INTERVENTIONS:
Device: functional Magnetic Resonance Imaging — In a 2-hour session, the subject we be shown different control and experimental conditions (all being visual stimuli) in perceptive tasks.

SUMMARY:
Little is known about the exact role of feedback in cortical processing. Hypotheses on its function range from attentional control to the transmission of Bayesian priors in the interpretation of sensory events, such as in the theory of Predictive Coding. Recent advances in identification of functional signatures of feedback and feedforward signal, as well as additional techniques based on causal relations in signal processing open a unique methodology for probing such processes in awake and behaving organisms and testing these theories and more generally the hierarchical processing between cortical areas.

The objective of this project is to study feedback and feedforward relations and localization in the well established pathways between cortical areas V1 and Medial Temporal (MT) that have been implicated in early integration processes in motion perception.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 40 years old
* Affiliated to a social security scheme
* Be right-handed
* Have signed the informed consent

Exclusion Criteria:

* Subjects with a neurological or psychiatric history
* Subjects with visual disturbances not corrected
* Pregnant, lactating or childbearing women without contraception.
* Persons under guardianship, trusteeship or any other administrative or judicial measure of deprivation of rights or liberty, as well as adults protected by law.
* Participants refusing to be informed of the results of the medical examination.
* Participants refusing to be informed of the possible detection of an anomaly.
* Volunteers with contraindications to the MRI examination: people using a pacemaker or an insulin pump, persons wearing a metal prosthesis or an intracerebral clip as well as claustrophobic subjects, neurosensory stimulator or implantable defibrillator, cochlear implants, ferromagnetic foreign body ocular or cerebral close to the nerve structures, agitation of the subject (non-cooperating or agitated subjects), ventriculoperitoneal neurosurgical bypass valves, dental apparatus.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07-22 (Actual); Primary Completion 2021-02-17 (Actual); Study Completion 2021-02-17 (Actual)

PRIMARY OUTCOMES:
Non-invasive Blood oxygenation level dependent (BOLD) fMRI activity | At inclusion
  Blood oxygenation level dependent (BOLD) imaging is the standard technique used to generate images in fMRI studies, and relies on regional differences in cerebral blood flow to delineate regional activity. This non-invasive technic is not inducing any particular risk. The non invasive BOLD fMRI activity will be recorded in healthy subjects during a task of visual perception.